CLINICAL TRIAL: NCT06377969
Title: Prospective Evaluation of Effectiveness and Safety of Closed-Loop Spinal Cord Stimulation in Treating Patients With Chronic Pelvic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vafi Salmasi, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 75269
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pelvic Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Pilot prospective single arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Patient will go through trial of spinal cord stimulator. If trial results in >50% reduction in pain, they will receive implantable spinal cord stimulator
  Interventions: Device: ECAP (Evoked Compound Action Potential)-controlled Closed-Loop Spinal Cord Stimulation

INTERVENTIONS:
Device: ECAP (Evoked Compound Action Potential)-controlled Closed-Loop Spinal Cord Stimulation — The patients will receive externalized epidural leads connected to external pulse generator for 5-14 days during trial phase. If the trial results in >50% reduction in pain, they will undergo a minor surgery to receive implantable spinal cord stimulator

SUMMARY:
Spinal cord stimulation (SCS) is an effective treatment for patients with chronic pelvic pain. The investigators will evaluate how safe and effective closed-loop spinal cord stimulation is in treating these patients; closed-loop spinal cord stimulation is a more novel method in delivering spinal cord stimulation that controls energy output of the device based on real-time feedback on how the device is stimulating the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include all adult patients (18 or older) with pelvic pain more than 6 months that has not responded to conservative medical management

Exclusion Criteria:

* Major untreated medical comorbidities (uncontrolled diabetes mellitus, severe obesity, uncontrolled cardiopulmonary disease, etc.)
* Secondary causes of pelvic pain that can be treated with appropriate medical or surgical interventions
* Major untreated psychological comorbidities
* Anatomical challeneges to place spinal cord stimulator
* Ongoing legal or disability claims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline, 3-month, 6-month and 12-month
  Numerical Rating Scale (0-10; higher score is worse)

SECONDARY OUTCOMES:
Change in Disability | Baseline, 3-month, 6-month and 12-month
  Pain Disability Index
Patient Global Impression Change | Baseline, 3-month, 6-month and 12-month
  7-point Likert Scale
Change in Quality of Life | Baseline, 3-month, 6-month and 12-month
  Short Form McGill Pain Questionnaire
Change in Pain Catastrophizing Scale | Baseline, 3-month, 6-month and 12-month
  14-item questionnaire scoring 0-52 (higher score worse)
Change in sleep quality | Baseline, 3-month, 6-month and 12-month
  PROMIS (Patient Reported Outcomes Measure Information System) Sleep Disturbance (t-score and percentile)
Change in Social Functioning | Baseline, 3-month, 6-month and 12-month
  PROMIS Satisfaction with social roles and activities (t-score and percentile)

IPD SHARING:
Plan to Share IPD: No